CLINICAL TRIAL: NCT04011267
Title: Effect of Customized Software for Foot-related Exercises (SOPeD) for Prevention and Treatment of Foot Musculoskeletal Dysfunctions of People With Diabetic Neuropathy: FOotCAre (FOCAtrial-I) Randomized Controlled Trial
Brief Title: Effect of Customized Software for Foot-related Exercises (SOPeD) for Prevention and Treatment in People With Diabetic Neuropathy
Acronym: FOCA-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Isabel de Camargo Neves Sacco, Associate Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FOCA-I
Record Dates: First submitted 2019-06-11; First posted 2019-07-08 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Diabetic Neuropathies
Keywords: exercise therapy; diabetic foot; preventive care; foot-related exercises; self-management; software; musculoskeletal function
MeSH Terms: conditions — Diabetic Neuropathies; Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients in the intervention group will perform foot-related exercises described in the SOPeD software three times/week at home via web-software. In the follow-up period, patients will follow the same schedule set by the project till the end of the study.
  Interventions: Other: Physical therapy by foot-ankle segmental and functional exercises
- Control Group (No Intervention): Participants in the control group will not receive any specific intervention in addition to the treatment recommended by the health professionals team (doctors, nurses, podiatrists), which includes pharmacological treatment, and self-care recommendations and foot care by international consensus.

INTERVENTIONS:
Other: Physical therapy by foot-ankle segmental and functional exercises — The physiotherapeutic foot-ankle exercise protocol is based on previous clinical trials. It was designed following three criteria established in a supervised, face-to-face intervention: muscle stretching; strengthening of the intrinsic muscles; and strengthening of the extrinsic foot-ankle muscles and functional exercises, such as balance and gait training. To avoid monotony, game principles were inserted to reward the exercise execution and enhance motivation. The exercises change from session to session, and the maximum duration is no longer than 20 minutes. The exercises should only be done 3 times/week; no more than eight exercises each day; and the individual difficulty is regulated by the effort scale to manage the customized progression. In total, 39 different exercises were chosen, and when including their sublevels of progression, a total of 104 different exercises can be completed.
  Arms: Intervention Group

SUMMARY:
The main objective of this trial is to investigate the effect of a customized foot-related exercises software (SOPeD) in diabetic neuropathy status, functional outcomes and gait biomechanics in people with diabetic neuropathy.

DETAILED DESCRIPTION:
A randomized controlled trial will be performed with 62 patients with diabetic neuropathy. The participants will be randomly assigned into either a control group (recommended foot care by international consensus with no foot exercises) or an intervention group that will perform exercises at home, three times a week, through the SOPeD (Diabetic Foot Guidance System) software for 12-weeks. The exercise program is customized during the performance by a perceived effort scale reported by the participant.

The subjects will be evaluated in 3 different times to access the effect of the intervention: baseline and 12 weeks, for all outcomes; and 24 weeks, for follow-up reasons for all outcomes. The following outcomes will be assessed in all times: (1) diabetic neuropathy symptoms and signs by Michigan Neuropathy Screening Instrument, (2) fuzzy score of the neuropathy severity, (3) foot-ankle kinematics during gait (infrared cameras) (4) foot-ankle joint moment during gait (infrared cameras and force plate), (5) plantar pressure distribution during gait, (6) tactile (monofilaments), (7) vibration sensitivity (tuning fork), (8) foot health and functionality by the Foot Health Status Questionnaire, (9) Foot isometric strength (pressure plate measurement), (10) functional balance reach test.

The hypothesis of this study is that the intervention will increase the perception of the tactile and vibratory sensitivity of the foot, reduce the symptoms of diabetic neuropathy, increase the strength of the foot muscles, increase the functional balance score, decrease the severity of the diabetic neuropathy (fuzzy score), decrease the number of neuropathy symptoms, promote a more physiological foot rollover with a redistribution of plantar pressure during gait, as well as increase foot-ankle mobility after 12-weeks of intervention. There will be also beneficial biomechanical changes during gait, such as: (1) increase in the ankle extensor moment and ankle concentric power in the propulsion phase and (3) increase in the ankle flexor moment and ankle eccentric power in the load phase.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 1 or 2;
* Moderate or severe neuropathy confirmed with the fuzzy software;
* Ability to walk independently in the laboratory ;
* Accessibility to electronic devices (computers, mobile devices, tablets, etc.) access to exercise software.

Exclusion Criteria:

* Hallux amputation or total amputation of the foot;
* History of surgical procedure in the knee, ankle or hip;
* History of arthroplasty and / or lower limb orthosis or indication of lower limb arthroplasty throughout the intervention period;
* Neurological and / or rheumatologic diseases diagnosed;
* Inability to provide consistent information;
* Perform physiotherapy intervention throughout the intervention period;
* Receiving any physiotherapy intervention or offloading devices;
* Major vascular complications;
* Severe retinopathy;
* Ulceration not healed for at least 6 months and / or active ulcer;
* Score between 12-21 (Probable Depression) from the Hospital Anxiety and Depression Scale (HADS).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Diabetic neuropathy symptoms at 12-weeks | 12-weeks, 24-weeks (follow-up)
  Score of the Michigan Neuropathy Screening Instrument (MNSI). This questionnaire comprises 15 questions about symptoms and events related to leg and foot sensitivity and is administered by the participant himself. The answers are summed to get a total score. The sum of all items results in a score ranging from 0 to 13 (13 represents the worst rating of the diabetic neuropathy).
Change from Baseline of the Fuzzy classification of the diabetic neuropathy severity at 12-weeks | 12-weeks, 24-weeks (follow-up)
  The fuzzy classification of the diabetic neuropathy severity will be given by the Fuzzy software score developed by the Laboratory of Biomechanics of Movement and Human Posture, available free of charge at: http://www.usp.br/labimph/fuzzy/. It is a decision support system for classification of the diabetic neuropathy. This decision is based on three domains: signs and symptoms extracted from the Michigan Neuropathy Screening Instrument; tactile sensitivity through the number of non-sensible areas using a 10-g monofilament; and vibration sensitivity by vibrating a tuning fork (128Hz) characterized as absent, present or diminished. The software produces a score from 0 to 10 and the higher the score, the more severe the diabetic neuropathy.

SECONDARY OUTCOMES:
Change from Baseline of the foot and ankle kinematics during gait at 12-weeks | 12-weeks, 24-weeks (follow-up)
  Ankle & Foot joints and plantar arch motion: maximum, minimum and range of motion (degrees) during gait
Change from Baseline of the foot-ankle joint moment during gait at 12-weeks | 12-weeks, 24-weeks (follow-up)
  maximum foot-ankle joint moment (joint loads N.m), calculated by inverse dynamics during gait.
Change from Baseline Dynamic Plantar Pressure Distribution during gait at 12-weeks | 12-weeks, 24-weeks (follow-up)
  A pressure platform (emed®-q100, novel, Germany) will be used to evaluate the pressure pattern during walking. The analysis of plantar pressure will be through the parameters: peak pressure (kPa), pressure - time integral (kPa/s) in each plantar area.
Change from Baseline Tactile sensitivity at 12-weeks | 12-weeks, 24-weeks (follow-up)
  Tactile sensorial deficits will be evaluated by monofilament with a tactile stimulus of a 10-g monofilament in 4 plantar areas (plantar face of the hallux, heads of 1st, 3rd and 5th metatarsals). The areas will be evaluated in random order and not allowing the participant to view the monofilament. The number of areas where the participant does not feel the pressure will be indicated. The greater the number of areas marked without sensing, the greater the impairment of tactile sensitivity.
Change from Baseline Vibration sensitivity at 12-weeks | 12-weeks, 24-weeks (follow-up)
  The vibration sensitivity will be assessed by vibrating a tuning fork (128Hz) in the dorsal region of the distal hallux phalanx. The participant should report the moment he/she does no longer feel the vibration of the tuning fork, and the evaluator must time the interval between which the participant reports that he/she ceases to feel the vibration and the moment the evaluator ceases to feel the vibration in the his/her hand. Values smaller than 10 seconds will be classified with present vibratory sensitivity; values greater than 10 seconds will be classified as decreased vibratory sensitivity. If the participant does not perceive the vibration imposed by the tuning fork, it will be classified as absent vibratory sensitivity.
Change from Baseline Foot health and functionality at 12-weeks | 12-weeks, 24-weeks (follow-up)
  The Brazilian version of the Foot-Health Status Questionnaire (FHSQ-BR) will be used. This instrument is divided into three domains and we are using domains I and II. The first domain evaluates the foot in four spheres: pain, function, footwear and general health. The second domain evaluates the general state of health, also in four spheres: general health, physical activity, social capacity and vitality. Domains I and II are composed of questions with answer choices that are presented in the affirmative sentences and corresponding numbers. Domain III, which is not being used, comprises the collection of general demographic data of individuals. Each domain receives a score from 0 to 100, where 100 expresses the best condition and 0 to worst.
Change from Baseline Foot isometric strength at 12-weeks | 12-weeks, 24-weeks (follow-up)
  The muscle strength of the flexor muscles of the hallux and flexors of the toes will be evaluated using the emed®-q100 pressure platform (novel, Germany) according to a test protocol already described elsewhere. The individual should stand, with the evaluated foot centered on the pressure platform, instructed to make as much force as possible with the hallux and toes in order to press them against the platform ("squeeze the platform with the toes"). Peak values of maximum force (N) will be extracted. The values will be normalized by bodyweight.
Change from Baseline Functional balance at 12-weeks | 12-weeks, 24-weeks (follow-up)
  It is a clinical test where the patient will be standing barefoot, perpendicular to the wall, with the shoulder flexed 90° and the elbow extended. A tape measure will be attached to the wall, parallel to the floor, positioned at the height of the patient's acromion. The volunteer will be instructed to lean forward as much as possible without losing balance or taking a step. The displacement of the wrist will be measured by the tape. The greater the distance in centimeter, the better the functional balance.
Cost Effectiveness and cost utility | 12-weeks, 24-weeks (follow-up)
  Assessments of costs by an specific questionnaire and the database of the public health system
Quality Adjusted Life Years | 12-weeks, 24-weeks (follow-up)
  Quality adjusted life years will be measured by the EQ-5D-3L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Isabel de Camargo Neves Sacco, PhD, Principal Investigator — Associate Professor at São Paulo University
Locations (1):
- Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferreira JSSP, Cruvinel-Junior RH, da Silva EQ, Verissimo JL, Monteiro RL, Duarte M, Giacomozzi C, Sacco ICN. Effectiveness of a web-based foot-ankle exercise program for treating ulcer risk factors in diabetic neuropathy in a randomized controlled trial. Sci Rep. 2024 Nov 8;14(1):27291. doi: 10.1038/s41598-024-78188-7. PMID 39516524
- [Derived] Cruvinel-Junior RH, Ferreira JSSP, Verissimo JL, Monteiro RL, Silva EQ, Suda EY, Sacco ICN. Affordable web-based foot-ankle exercise program proves effective for diabetic foot care in a randomized controlled trial with economic evaluation. Sci Rep. 2024 Jul 12;14(1):16094. doi: 10.1038/s41598-024-67176-6. PMID 38997439
- [Derived] Cruvinel Junior RH, Ferreira JSSP, Beteli RI, Silva EQ, Verissimo JL, Monteiro RL, Suda EY, Sacco ICN. Foot-ankle functional outcomes of using the Diabetic Foot Guidance System (SOPeD) for people with diabetic neuropathy: a feasibility study for the single-blind randomized controlled FOotCAre (FOCA) trial I. Pilot Feasibility Stud. 2021 Mar 26;7(1):87. doi: 10.1186/s40814-021-00826-y. PMID 33766146
- [Derived] Ferreira JSSP, Cruvinel Junior RH, Silva EQ, Verissimo JL, Monteiro RL, Pereira DS, Suda EY, Sartor CD, Sacco ICN. Study protocol for a randomized controlled trial on the effect of the Diabetic Foot Guidance System (SOPeD) for the prevention and treatment of foot musculoskeletal dysfunctions in people with diabetic neuropathy: the FOotCAre (FOCA) trial I. Trials. 2020 Jan 13;21(1):73. doi: 10.1186/s13063-019-4017-9. PMID 31931855
- See also: University of Sao Paulo website — http://www.usp.br
- See also: Laboratory of Biomechanics of Human Movement and Posture website — http://www.usp.br/labimph
- See also: Educational Diabetic Foot Software — http://www.soped.com.br